CLINICAL TRIAL: NCT02364947
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, 3-parallel-group Comparison Trial to Investigate the Effect of Nalmefene on Alcohol Consumption Reduction in Patients With Alcohol Dependence (Phase 3 Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 339-14-001; JapicCTI-152804 (Other: Japic)
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-07

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — nalmefene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nalmefene hydrochloride 10 mg (Experimental)
  Interventions: Drug: Nalmefene hydrochloride
- Nalmefene hydrochloride 20 mg (Experimental)
  Interventions: Drug: Nalmefene hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nalmefene hydrochloride — As-needed; tablets, orally
  Arms: Nalmefene hydrochloride 10 mg; Nalmefene hydrochloride 20 mg
Drug: Placebo — As-needed; tablets, orally
  Arms: Placebo

SUMMARY:
The efficacy, safety, and dose-response of nalmefene hydrochloride at 10 mg and 20 mg in patients with alcohol dependence will be evaluated in a multicenter, randomized, double-blind, placebo-controlled, 3-parallel-group comparative trial. The superiority of nalmefene hydrochloride at 20 mg to placebo will be verified in terms of reduction of alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* Japanese males and females aged 20 or above who have signed the informed consent form
* The patient has alcohol dependence, diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) and confirmed by Mini-international Neuropsychiatric Interview (M. I. N. I.)
* The patient has a drinking risk level of High or above (> 60 g for men and > 40 g for women) both at the Screening Visit and at the Randomization Visit .

Exclusion Criteria:

* The patient with a current diagnosis or history of substance use disorders (except for alcohol, nicotine, and caffeine), according to DSM-IV-TR and confirmed by M. I. N. I.
* The patient has reported current use of, or has tested positive for, drugs of abuse (opiates, methadone, cocaine, amphetamines, barbiturates) at the screening test

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2015-02-09 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Sato, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (7):
- Japan (7):
  - Chubu, Region
  - Hokkaido, Region
  - Kanto, Region
  - Kinki, Region
  - Kyusyu, Region
  - Tohoku, Region
  - Tyugoku, Region

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Safety analysis set, which included all randomized patients who received ≥1 dose of the study medication.
Groups:
- Nalmefene Hydrochloride 20 mg; Nalmefene Hydrochloride 10 mg; Placebo: as-needed, tablets, orally, 24 weeks
Period: Overall Study
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Started | 248 | 184 | 245
Completed | 189 | 139 | 219
Not Completed | 59 | 45 | 26
Not completed — Withdrawal by Subject | 10 | 8 | 9
Not completed — Adverse Event | 45 | 33 | 11
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Physician Decision | 3 | 2 | 5
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo | Total
Number analyzed (Participants) | 242 | 180 | 244 | 666
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 213 | 159 | 217 | 589
  >=65 years | 29 | 21 | 27 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (12.2) | 49.2 (11.9) | 48.1 (11.4) | 48.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 46 | 90 | 208
  Male | 170 | 134 | 154 | 458
Region of Enrollment [Number; unit: participants]
  Japan | 242 | 180 | 244 | 666
Heavy Drinking Days (HDDs) [Mean (Standard Deviation); unit: days/month] — The number of HDDs was defined as the number of days per month [days/month] with alcohol consumption of > 60 g for males and > 40 g for females.
  days/month | 22.64 (6.37) | 23.49 (6.07) | 22.97 (6.44) | 22.99 (6.32)
Total Alcohol Consumption (TAC) [Mean (Standard Deviation); unit: g/day] — TAC was defined as mean alcohol consumption per day [g/day] over a 1-month period.
  g/day | 93.07 (37.45) | 95.93 (41.10) | 95.08 (48.70) | 94.58 (42.79)
Drinking Risk Level (DRL) [Count of Participants; unit: Participants] — DRL was defined by the World Health Organization based on average volume of alcohol consumption per Day.
  Participants
    Low | 0 | 0 | 0 | 0
    Medium | 0 | 0 | 1 | 1
    High | 135 | 93 | 127 | 355
    Very high | 107 | 87 | 116 | 310
Clinical Global Impression - Severity of Illness (CGI-S) score [Mean (Standard Deviation); unit: units on a scale] — The CGI-S scale was used by clinicians when assessing their global impression of a patient's current clinical condition. The investigator or subinvestigator used his/her clinical experience with this patient population to rate the severity of a subject's clinical condition on a 7-point scale ranging from 1 (Normal, not at all ill) to 7 (Among the most extremely ill patients).
  units on a scale | 3.38 (1.06) | 3.48 (1.15) | 3.45 (1.09) | 3.43 (1.09)
Serum gamma-glutamyltransferase (γ-GT) [Mean (Standard Deviation); unit: IU/L] | 84.7 (105.4) | 80.7 (103.8) | 70.7 (78.7) | 78.5 (96.1)
Serum alanine aminotransferase (ALT) [Mean (Standard Deviation); unit: IU/L] | 24.3 (14.2) | 24.5 (14.9) | 23.3 (14.8) | 24.0 (14.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Heavy Drinking Days (HDDs) From Baseline at Week 12
Description: The number of HDDs is defined as the number of days per month [days/month] with alcohol consumption of > 60 g for males and > 40 g for females
Time Frame: Week 12
Population: Full analysis set, which included all patients who had data on the number of HDDs at baseline and at ≥1 time point after initiation of the study drug.
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
days/month | -12.25 (0.64) | -12.09 (0.74) | -7.91 (0.61)
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — Mixed model for repeated measures (MMRM) with fixed effect of treatment, sex, time point, treatment-by-time point interaction, baseline value, and baseline value-by-time point interaction with an unstructured variance-covariance matrix structure was used; p = 0.0001, Mixed Models Analysis — Efficacy of the doses (change from baseline in the number of HDDs vs placebo) was assessed using a closed testing procedure. The 20 mg dose was tested at a 5% level of significance and only if significant, the testing would proceed to the 10 mg dose; Mean Difference (Final Values) = -4.34, 95% CI 2-sided [-6.05 to -2.62], Standard Error of Mean 0.87
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.18, 95% CI 2-sided [-6.05 to -2.32], Standard Error of Mean 0.95

2. Secondary Outcome: Change in the Number of Heavy Drinking Days (HDDs) From Baseline at Week 24
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
days/month | -13.25 (0.66) | -13.88 (0.77) | -9.33 (0.63)
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.92, 95% CI 2-sided [-5.69 to -2.16], Standard Error of Mean 0.90
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -4.54, 95% CI 2-sided [-6.46 to -2.63], Standard Error of Mean 0.98

3. Secondary Outcome: Change in Total Alcohol Consumption (TAC) From Baseline at Week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: g/day
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
g/day | -44.90 (2.01) | -45.36 (2.32) | -32.43 (1.91)
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Change in total alcohol consumption (TAC) from baseline at Week 12; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -12.47, 95% CI 2-sided [-17.81 to -7.13], Standard Error of Mean 2.72
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -12.94, 95% CI 2-sided [-18.72 to -7.15], Standard Error of Mean 2.95

4. Secondary Outcome: Change in Total Alcohol Consumption (TAC) From Baseline at Week 24
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: g/day
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
g/day | -49.43 (2.13) | -49.55 (2.45) | -38.28 (1.99)
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -11.15, 95% CI 2-sided [-16.77 to -5.53], Standard Error of Mean 2.86
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = -11.27, 95% CI 2-sided [-17.37 to -5.17], Standard Error of Mean 3.11

5. Secondary Outcome: Response Shift Drinking Risk Level (RSDRL) at Week 12
Description: Proportion of patients with a downward shift in drinking risk level of two categories or more
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
percentage | 41.3 | 35.7 | 20.1
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline DRL; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 22.0, 95% CI 2-sided [13.6 to 30.4]
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline DRL; p = 0.0007, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.7, 95% CI 2-sided [6.5 to 25.0]

6. Secondary Outcome: Response Shift Drinking Risk Level (RSDRL) at Week 24
Description: Proportion of patients with a downward shift in drinking risk level of two categories or more
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
percentage | 44.4 | 47.5 | 27.5
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline DRL; p = 0.0002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 18.0, 95% CI 2-sided [8.8 to 27.2]
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline DRL; p = 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.6, 95% CI 2-sided [10.4 to 30.8]

7. Secondary Outcome: Response Low Drinking Risk Level (RLDRL) at Week 12
Description: Proportion of patients with low or lower drinking risk level
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
percentage | 29.6 | 25.3 | 10.7
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline DRL; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.8, 95% CI 2-sided [10.5 to 25.1]
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline DRL; p = 0.0002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 14.3, 95% CI 2-sided [6.4 to 22.2]

8. Secondary Outcome: Response Low Drinking Risk Level (RLDRL) at Week 24
Description: Proportion of patients with low or lower drinking risk level
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
percentage | 29.6 | 32.6 | 17.6
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline DRL; p = 0.0079, Cochran-Mantel-Haenszel; Risk Difference (RD) = 11.0, 95% CI 2-sided [2.9 to 19.1]
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline DRL; p = 0.0010, Cochran-Mantel-Haenszel; Risk Difference (RD) = 14.8, 95% CI 2-sided [5.8 to 23.9]

9. Secondary Outcome: 70% TAC Responder Rate at Week 12
Description: Proportion of patients with a 70% decrease in TAC
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
percentage | 18.0 | 19.5 | 8.5
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline value; p = 0.0022, Cochran-Mantel-Haenszel; Risk Difference (RD) = 9.9, 95% CI 2-sided [3.5 to 16.3]
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline value; p = 0.0016, Cochran-Mantel-Haenszel; Risk Difference (RD) = 11.1, 95% CI 2-sided [3.8 to 18.3]

10. Secondary Outcome: 70% TAC Responder Rate at Week 24
Description: Proportion of patients with a 70% decrease in TAC
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
percentage | 23.8 | 23.4 | 10.8
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline value; p = 0.0003, Cochran-Mantel-Haenszel; Risk Difference (RD) = 13.6, 95% CI 2-sided [6.2 to 20.9]
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline value; p = 0.0013, Cochran-Mantel-Haenszel; Risk Difference (RD) = 12.8, 95% CI 2-sided [4.6 to 21.0]

11. Secondary Outcome: HDD Responder Rate at Week 12
Description: Proportion of patients with ≤4 HDDs
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
percentage | 35.0 | 36.4 | 19.2
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline value; p = 0.0002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.2, 95% CI 2-sided [7.1 to 23.3]
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline value; p = 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.9, 95% CI 2-sided [8.9 to 26.9]

12. Secondary Outcome: HDD Responder Rate at Week 24
Description: Proportion of patients with ≤4 HDDs
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
percentage | 33.9 | 44.0 | 25.2
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline value; p = 0.0724, Cochran-Mantel-Haenszel; Risk Difference (RD) = 8.0, 95% CI 2-sided [-0.7 to 16.7]
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — Cochran-Mantel-Haenszel test, stratified by sex and baseline value; p = 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 19.6, 95% CI 2-sided [9.9 to 29.2]

13. Secondary Outcome: Change in CGI-S From Baseline at Week 12
Description: The CGI-S scale was used by clinicians when assessing their global impression of a patient's current clinical condition. The investigator or subinvestigator used his/her clinical experience with this patient population to rate the severity of a subject's clinical condition on a 7-point scale ranging from 1 (Normal, not at all ill) to 7 (Among the most extremely ill patients).
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
units on a scale | -0.60 (0.05) | -0.63 (0.06) | -0.34 (0.05)
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.40 to -0.13], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.45 to -0.15], Standard Error of Mean 0.08

14. Secondary Outcome: Change in CGI-S From Baseline at Week 24
Description: as for outcome 13
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
units on a scale | -0.75 (0.06) | -0.77 (0.07) | -0.41 (0.05)
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.48 to -0.18], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.51 to -0.19], Standard Error of Mean 0.08

15. Secondary Outcome: Change in CGI-I From Baseline at Week 12
Description: The CGI-I scale is used to assess a patient's improvement (or worsening). The investigator or subinvestigator assesses a subject's condition relative to baseline on a 7-point scale ranging from 1 (Very much improved) to 7 (Very much worse).
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
units on a scale | 2.62 (0.07) | 2.65 (0.08) | 3.13 (0.06)
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — Mixed model for repeated measures (MMRM) with fixed effect of treatment, sex, time point, treatment-by-time point interaction, baseline value, and baseline value-by-time point interaction with an unstructured variance-covariance matrix structure was used. Baseline CGI-S value was used as baseline value in MMRM; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.69 to -0.33], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 15, analysis 1]; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.67 to -0.27], Standard Error of Mean 0.10

16. Secondary Outcome: Change in CGI-I From Baseline at Week 24
Description: The CGI-I scale was used to assess a patient's improvement (or worsening). The investigator or subinvestigator assesses a subject's condition relative to baseline on a 7-point scale ranging from 1 (Very much improved) to 7 (Very much worse).
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
units on a scale | 2.49 (0.07) | 2.44 (0.09) | 2.99 (0.07)
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 15, analysis 1]; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.70 to -0.31], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 15, analysis 1]; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.77 to -0.33], Standard Error of Mean 0.11

17. Secondary Outcome: Change in Logarithm Scale in Serum γ-glutamyltransferase From Baseline at Week 12
Description: All-patients-randomised set
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
IU/L | 3.666 (0.027) | 3.702 (0.031) | 3.858 (0.025)
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — Mixed model for repeated measures (MMRM) with fixed effect of treatment, sex, time point, treatment-by-time point interaction, logarithm scale baseline value, and logarithm scale baseline value-by-time point interaction with an unstructured variance-covariance matrix structure was used; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.192, 95% CI 2-sided [-0.262 to -0.121], Standard Error of Mean 0.036
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 17, analysis 1]; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.156, 95% CI 2-sided [-0.232 to -0.080], Standard Error of Mean 0.039

18. Secondary Outcome: Change in Logarithm Scale in Serum γ-glutamyltransferase From Baseline at Week 24
Description: All-patients-randomised set
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
IU/L | 3.663 (0.031) | 3.692 (0.035) | 3.831 (0.028)
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 17, analysis 1]; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.168, 95% CI 2-sided [-0.248 to -0.088], Standard Error of Mean 0.041
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 17, analysis 1]; p = 0.0017, Mixed Models Analysis; Mean Difference (Final Values) = -0.139, 95% CI 2-sided [-0.226 to -0.052], Standard Error of Mean 0.044

19. Secondary Outcome: Change in Logarithm Scale in Serum Alanine Aminotransferase From Baseline at Week 12
Description: All-patients-randomised set
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
IU/L | 2.968 (0.023) | 2.988 (0.027) | 3.038 (0.021)
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 17, analysis 1]; p = 0.0234, Mixed Models Analysis; Mean Difference (Final Values) = -0.070, 95% CI 2-sided [-0.130 to -0.009], Standard Error of Mean 0.031
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Mixed model for repeated measures (MMRM) with fixed effect of treatment, sex, time point, treatment-by-time point interaction, logarithm scale baseline value, and logarithm scale baseline value-by-time point interaction with an unstructured variance-covariance matrix structure was used; Test type: Superiority or Other; p = 0.1374, Mixed Models Analysis; Mean Difference (Final Values) = -0.049, 95% CI 2-sided [-0.115 to 0.016], Standard Error of Mean 0.033

20. Secondary Outcome: Change in Logarithm Scale in Serum Alanine Aminotransferase From Baseline at Week 24
Description: All-patients-randomised set
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
Number analyzed (Participants) | 242 | 180 | 244
IU/L | 2.971 (0.023) | 2.987 (0.027) | 3.036 (0.021)
Statistical Analysis 1: Comparison: Nalmefene Hydrochloride 20 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 17, analysis 1]; p = 0.0348, Mixed Models Analysis; Mean Difference (Final Values) = -0.066, 95% CI 2-sided [-0.127 to -0.005], Standard Error of Mean 0.031
Statistical Analysis 2: Comparison: Nalmefene Hydrochloride 10 mg vs Placebo; Test type: Superiority or Other — [test comment as in outcome 17, analysis 1]; p = 0.1444, Mixed Models Analysis; Mean Difference (Final Values) = -0.049, 95% CI 2-sided [-0.116 to 0.017], Standard Error of Mean 0.034

ADVERSE EVENTS:
Time Frame: 24-week treatment period
Arm/Group | Nalmefene Hydrochloride 20 mg | Nalmefene Hydrochloride 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/248 | 1/184 | 0/245
Serious Adverse Events (participants affected / at risk) | 2/248 | 2/184 | 2/245
Other Adverse Events (participants affected / at risk) | 175/248 | 125/184 | 127/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nalmefene Hydrochloride 20 mg (N=248) | Nalmefene Hydrochloride 10 mg (N=184) | Placebo (N=245)
Chronic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nalmefene Hydrochloride 20 mg (N=248) | Nalmefene Hydrochloride 10 mg (N=184) | Placebo (N=245)
Palpitations (Cardiac disorders) | 13 | 7 | 2
Constipation (Gastrointestinal disorders) | 13 | 8 | 2
Nausea (Gastrointestinal disorders) | 79 | 58 | 15
Vomiting (Gastrointestinal disorders) | 34 | 16 | 5
Malaise (General disorders) | 24 | 7 | 8
Nasopharyngitis (Infections and infestations) | 54 | 40 | 91
Decreased appetite (Metabolism and nutrition disorders) | 13 | 11 | 3
Dizziness (Nervous system disorders) | 51 | 20 | 10
Headache (Nervous system disorders) | 24 | 21 | 20
Somnolence (Nervous system disorders) | 39 | 18 | 17
Insomnia (Psychiatric disorders) | 20 | 15 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No